CLINICAL TRIAL: NCT03069534
Title: Study of Adjunctive rhIL-2 Therapy in Patients With MDR-TB That Improves Efficiency and Shortens Course
Brief Title: Study of Adjunctive Recombinant Human Interleukin-2 Therapy in Patients With MDR-TB
Acronym: rhIL-2
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rhIL-2 Therapy ON MDR-TB
Record Dates: First submitted 2017-02-19; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2009-09

CONDITIONS: MDR TB
Keywords: MDR-TB; rhIL-2; immunotherapy
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rhIL-2 Group (Experimental): The patients in rhIL-2 Group were given consisted of four courses of low-dose rhIL-2 plus standard anti-tuberculosis chemotherapy. rhIL-2 (500，000U/m)regiman was given subcutaneously (SC) once every other day (q.o.d.) for 30 days and four courses were carried out separately during months 1, 3, 5, and 7. Standard anti-MDR-TB chemotherapy regiman was totally 24 months,including 6-month Z+KM/AM or CM + PAS/(Pa) + PTO +LFX as an intensive phase treatment, followed by an 18-month Z + LFX + PTO + PAS/(Pa) as a consolidation phase treatment.Then all the group patients were followed up for a minimum of 36 months.
  Interventions: Drug: RhIL-2
- Control Group (No Intervention): The patients in Control Group were given standard anti-tuberculosis chemotherapy regiman.Standard anti-MDR-TB chemotherapy regiman was totally 24 months,including 6-month Z+KM/AM or CM + PAS/(Pa) + PTO +LFX as an intensive phase treatment, followed by an 18-month Z + LFX + PTO + PAS/(Pa) as a consolidation phase treatment.Then all the group patients were followed up for a minimum of 36 months

INTERVENTIONS:
Drug: RhIL-2 — RhIL-2 treatment intervention was consisted of four courses of low-dose rhIL-2 plus standard anti-tuberculosis chemotharapy. rhIL-2 (500,000 U/m)regimen was given subcutaneously (SC) once every other day (q.o.d.) for 30 days and four courses were carried out separately during months 1, 3, 5, and 7.
  Arms: rhIL-2 Group

SUMMARY:
Multidrug-resistant tuberculosis (MDR-TB) has emerged as a challenge worldwide. Few studies have prospectively reported outcomes in patients with pulmonary MDR-TB treated with adjunctive immunotherapy combined to standard chemotherapy. We aimed to assess whether immunotherapy with Interleukin(IL)-2 enhanced the clinical and immune effects of treatment on MDR-TB patients.We performed a multicentre prospective cohort study extend all over Jiangsu province in China. Two groups were generated based on the adjunctive rhIL-2 therapy during 24 months regiman. Bacteriological and imaging data were followed during 24 months with cure rates analysed.

DETAILED DESCRIPTION:
IL-2 therapy regimans are expected to restore the immune response or to change the immunologic status,thus allowing the host to more efficiently contain and eradicate immune responses, primarily those against cancers and infectious diseases.To address this, we performed a prospective randomized controlled multicenter cohort study of 8-month adjunctive immunotherapy with rhIL-2 for MDR-TB patients compared with the standard chemotherapy.

This multicenter prospective clinical study was conducted at 13 tuberculosis centers (coordinating hospital specialized in tuberculosis) across Jiangsu province, China. Joined by the network system of The First Affiliated Hospital of Nanjing Medical University and CDC of Jiangsu province, participants were enrolled from 2009 to 2018. This study protocol was approved by the ethics committee of the First Affiliated Hospital of Nanjing Medical University and was performed adhering to the ethical principles of the Declaration of Helsinki. All patients provided written informed consent before enrollment. The independent data and safety of the study were monitored by the hospital monitoring committee.

Patients enrollment

Eligible MDR-TB participants were identified by triplicate-spot sputum smears that were positive for acid-fast bacilli and a positive sputum culture with resistance to both isoniazid and rifampin, as determined by susceptibility tests and rapid screening tests . The results of these assays were confirmed using an L-G medium base modified in the Jiangsu province Centers for Disease Control and Prevention（CDC）.

Treatment plan for the two cohorts: The patients in rhIL-2 group were given consisted of four courses of low-dose rhIL-2 (500，000 U/m) given subcutaneously (SC) once every other day (q.o.d.) for 30 days. Four courses were carried out separately during months 1, 3, 5, and 7. All enrolled patients with pulmonary MDR-TB received a 24-month standard anti-MDR-TB chemotherapy regimen:6-month Z+KM/AM or CM + PAS/(Pa) + PTO +LFX as an intensive phase treatment, followed by an 18-month Z + LFX + PTO + PAS/(Pa) as a consolidation phase treatment.

(Z: Pyrazinamide; KM: Kanamycin; AM: Amikacin; CM: Capreomycin; LFX: Levofloxacin; PTO: Prothionamide; PAS: Para-aminosalicylicacid; Pa:Pasiniazid); After finishing treatment regimen patients were followed up for a minimum of 36- months or until discontinuation of regimen, withdrawal of consent, loss to follow-up, death, or end of study.

For all of the participants demographic measurements were recorded on the first clinical visit. Patient data were collected at enrollment and quarterly intervals. Sputum smear conversion, sputum culture conversion and chest CT scan improvement were followed up at 3, 6, 12, 18, and 24 months for bacteriological and imaging data collected. Cure rates analysed and compared in both groups.

The proportions of MDR-TB patients in the two groups achieving sputum smear/culture conversion, lung lesions absorption were assessed and compared.

Safety assessment included clinical symptom observation, Incidences of adverse event （AE ）in two groups were assessed and compared. blood routine test, hematologic profile, blood biochemical examination including hepatic aminotransferase and blood ureantrogen/creatinine, blood electrolyte test (potassium, magnesium, calcium), serum thyroid stimulating hormone(TSH), audiology examinations, visual field and color examination.

Cure rate was defined as first outcome. Sputum conversion rate was defined as second outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients had/were:

1. a confirmed case of MDR-TB;
2. aged 18-70 years old;
3. a chest CT showing visible lung lesions, with or without holes;
4. a fasting plasma glucose of less than 7.8 mol/L and a normal fundus examination, if they were diabetic;
5. voluntarily joined this study and signed an informed consent form.

Exclusion Criteria:

1. two or more total allergies or any drug or food allergies;
2. resistant to some drugs of this program;
3. severe disorders of liver, kidney, or hematologic system functions;
4. any metabolic diseases, autoimmune diseases, endocrine diseases, cancer, or HIV/AIDS;
5. a long-term use of immunosuppressive agents;
6. a blood system dysfunction;
7. a history of mental illness or epilepsy;
8. pregnant or lactating;
9. participated in another clinical trial in the last 3 months or were currently participating in other ongoing clinical trials;
10. long-term alcohol abuse>10 years and more than two alcoholic drinks per day);
11. any other factor rendering them unsuitable to participate in this project, such as a history of unreliability.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate | 130 months
  Completion of treatment and at least five consecutive negative sputum cultures from samples collected at least 30 days apart or one positive sputum culture followed by a minimum of three consecutive negative cultures taken at least 30 days apart during the final 12 months of treatment;

SECONDARY OUTCOMES:
sputum smear/culture conversion rate | 24 months
  The proportions of MDR-TB patients in the two groups achieving sputum smear/culture conversion at the end of 24 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hong Wang, PH.D, Principal Investigator — the First Affiliated Hospital of Nanjing Medical University, Nanjing, China
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China